CLINICAL TRIAL: NCT04019691
Title: Comparing the Visual Outcome, Visual Quality, and Satisfaction Among Three Types of Multi-focal Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC 2019-06-017-001
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2020-04

CONDITIONS: Cataract
Keywords: multifocal intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mix-and-Match group (Active Comparator): Cataract surgery and implantation of a Tecnis ZKB00 multifocal IOL with +2.75 D add power (Abbott Medical Optic Inc., Santa Ana, CA) in the dominant eye, and a Tecnis ZLB00 multifocal IOL with +3.25 D add power (Abbott Medical Optics Inc.) in the non-dominant eye.
  Interventions: Device: Mix-and-Match
- EDOF group (Active Comparator): Cataract surgery and implantation of Tecnis Symfony ZXR00 trifocal IOLs (Abbot Medical Optics Inc.) in both eyes.
  Interventions: Device: EDOF
- Trifocal group (Active Comparator): Cataract surgery and implantation of FineVision PodFT IOLs (PhysIOL SA) in both eyes.
  Interventions: Device: Trifocal

INTERVENTIONS:
Device: Mix-and-Match — Phacoemulsification and implantation of Tecnis ZKB00 multifocal IOL with +2.75 D add power (Abbott Medical Optic Inc., Santa Ana, CA) in the dominant eye, and a Tecnis ZLB00 multifocal IOL with +3.25 D add power (Abbott Medical Optics Inc.) in the non-dominant eye.
  Arms: Mix-and-Match group
Device: EDOF — Phacoemulsification and implantation of Tecnis Symfony ZXR00 trifocal IOLs (Abbot Medical Optics Inc.) in both eyes.
  Arms: EDOF group
Device: Trifocal — Phacoemulsification and implantation of FineVision PodFT IOLs (PhysIOL SA) in both eyes.
  Arms: Trifocal group

SUMMARY:
The investigators are going to Investigate the comparative efficacy of the patients who underwent cataract surgery with three different multifocal IOLs.

DETAILED DESCRIPTION:
Going to analyze the clinical results of 60 patients who underwent bilateral cataract surgery and multifocal IOL implantation. The patients were divided into the following three groups: Mix-and-Match, EDOF, and Trifocal. The clinical assessments included uncorrected near, intermediate, distance and best corrected distance visual acuity, defocus curves, contrast sensitivity, and reading speed. Patient satisfaction was evaluated by questionnaire. All outcomes were compared among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral senile cataracts and the desire to be spectacle-free for all distances

Exclusion Criteria:

* Patients younger than 21 years, had corneal astigmatism >1.00 D, previous ocular surgery or trauma, or ocular disease other than cataracts

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Postoperative uncorrected near, intermediate, and far visual acuity. | At 1month and 3months after surgery
  logMAR
Postoperative contrast sensitivity in the three groups. | Postoperative 3 months
  3, 6, 12, and 18 cycles per degree using a CSV-1000 chart (Vector Vision, reenville, OH) under photopic (85 cd/m2), mesopic (~3 cd/m2), and mesopic with glare conditions
Postoperative satisfaction questionnaire. | Postoperative 3 months
  patients were shown images and asked to rate the frequency, degree, and discomfort related to the visual artifacts as none, minimal, moderate, or severe (0, 1, 2, or 3 points for the respective levels). The mean score was calculated.

SECONDARY OUTCOMES:
Postoperative refractive outcome | Postoperative 3 months
  Diopter

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paik DW, Park JS, Yang CM, Lim DH, Chung TY. Comparing the visual outcome, visual quality, and satisfaction among three types of multi-focal intraocular lenses. Sci Rep. 2020 Sep 9;10(1):14832. doi: 10.1038/s41598-020-69318-y. PMID 32908159